CLINICAL TRIAL: NCT03792412
Title: BagEL - Bariatric Patients in Primary Care: Post-operative Nutrition and Lifestyle Management Evaluation of a Post-operative Nutrition and Lifestyle Management for Lifelong Care of Post-bariatric Patients in Primary Care
Brief Title: BagEL - Bariatric Patients in Primary Care: Post-operative Nutrition and Lifestyle Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Krebs, Clinical Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2079/2017
Record Dates: First submitted 2018-12-01; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Bariatric Surgery Candidate; Malnutrition
Keywords: bariatric surgery; lifelong follow-up; primary care; obesity; health care study
MeSH Terms: conditions — Malnutrition; Obesity

STUDY DESIGN:
Intervention Model Description: randomised cohort study with control group
Who Masked: Participant
Masking Description: pseudonymity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Usability Questionnaire (Experimental): Patients hand over the usability questionnaire to evaluate the self developed structured follow-up program in form of a so-called pass to their family doctor twice in six months. Family doctors examine the postbariatric patient using the pass and evaluate the usability by filling out the questionnaire and return the usability questionnaire to the investigator.
  Interventions: Other: Usability Questionnaire
- Control: Usability Questionnaire (Other): Patients hand over the usability questionnaire to evaluate the state of the art guideline for postbariatric follow up appointments in form of a folder "Metabolische Chirurgie und die perioperative Betreuung" to their family doctor twice in six months. Family doctors examine the postbariatric patient using the guideline and evaluate the usability by filling out the questionnaire and return the usability questionnaire to the investigator.
  Interventions: Other: Usability Questionnaire

INTERVENTIONS:
Other: Usability Questionnaire — Patients receive the usability questionnaire and a structured nutrition and lifestyle program for post-bariatric follow-up visits. Twice in six months the patients visit their family doctor and hand over the usability questionnaire to evaluate the structured follow-up program for postbariatric patients. Family doctors fill out the questionnaire and returns it to the investigator.

SUMMARY:
There is a growing number of patients undergoing bariatric surgery requiring lifelong follow-up. BagEL (Bariatric Patients in Primary Care: Post-operative Nutrition and Lifestyle Management) is a survey to evaluate a newly developed structured disease management program including nutrition and lifestyle management in primary care.

DETAILED DESCRIPTION:
During last decades the prevalence of obesity is growing. Therefore, the number of bariatric procedures are also increasing. Frequent complications after surgery are nutritional deficiencies (e.g. vitamins, minerals, protein) which require mandatory long-term follow-up. So far adequate follow-up programs are only provided in specialized bariatric centers like in the outpatient clinic for obesity at the General Hospital of Vienna. These programs are focusing on prevention and premature identification of deficiencies.

Rising numbers of bariatric-surgical procedures pose a challenge for bariatric centres because of the accumulating numbers of bariatric patients requesting follow-up at least once a year.

To provide full coverage an appropriate possibility would be to transfer follow up to non-specialised facilities including general practitioners and family doctors using a so called "pass" providing practical treatment recommendations (necessary follow-up appointments, laboratory blood tests, questions regarding nutrition and lifestyle behavior).

To our best knowledge such a structured post-bariatric care management program in primary care does not exist by now. The aim of this study is therefore the evaluation of such a pass.

ELIGIBILITY:
Inclusion criteria:

* older than 18 years and each sex,
* bariatric-surgical treatment - in particular omega loop gastric bypass, Roux-en-Y-gastric bypass - and sleeve gastrectomy at the department of surgery General Hospital Vienna,
* Operation date maximum 21 months before study beginning,

Exclusion criteria:

* Pregnancy (a possible existing pregnancy is excluded by questioning)
* Nursing mothers
* Not German speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Usability questionnaire | 6 months
  Usability of the follow-up passes (intervention and control) will be evaluated in primary care. In a pilot study the usability questionnaire was evaluated.
  The patient hands over the follow-up pass together with the questionnaire at each appointment (twice) at the family doctor. A stamped envelope to return the questionnaire is included. Family doctors will be asked to complete a series of actions regarding the content of the follow-up passes. Each action will be rated in a 5 point likert scale. An average score will be calculated for each question.

SECONDARY OUTCOMES:
change in fat free mass | 6 months
  A Bioelectric impedance analysis will be used to calculate change in fat free mass. Measurements will be conducted by a device sending weak electric signals through the patients body. The method is non-invasive.
change in body weight | 6 months
  Patients will be asked to remove shoes, socks, heavy clothing and jewelry for measurement of body weight to the nearest 100 g using a digital scale.
Measures of adherence after 6 months | 6 months
  Number of patients returning to the outpatient clinic after the intervention.
Calcium Blood Value | 6 months
  Change in Calcium levels (mg/dL) after 6 months
Iron Blood Value | 6 months
  Change in Ferritin levels (ng/mL) after 6 months
Vitamin B12 Blood Value | 6 months
  Change in B12 levels (pmol/L) after 6 months
Vitamin D Blood Value | 6 months
  Change in Vitamin D, 25-Hydroxy levels (nmol/L) after 6 months
Folic Acid Blood Value | 6 months
  Change in Folic Acid levels (nmol/L) after 6 months
HbA1c Blood Value | 6 months
  Change in Hemoglobin A1c (%) after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Please Select, Austria